CLINICAL TRIAL: NCT03556735
Title: Evaluation Plan for Pulsed Electro Magnetic Fields (PEMF) in a Cohort Study for Patients With Unipolar Depression, Refractory to Antidepressant Drugs. A DUAG (Danish University Antidepressant Group) Study Over 8 Weeks.
Brief Title: Pulsed Electro Magnetic Fields (PEMF) in Depression
Acronym: PEMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Glostrup University Hospital, Copenhagen (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Erik Roj Larsen, Clinical associate professor, senior consultant, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-125-16
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2018-06

CONDITIONS: Depression, Unipolar
Keywords: Depression, unipolar; Treatment resistant; PEMF
MeSH Terms: conditions — Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEMF treatment (Other): No sham group (placebo) was chosen. Treatment consisted of one active group in a multicenter study.
  Interventions: Device: Treatment with PEMF equipment

INTERVENTIONS:
Device: Treatment with PEMF equipment — Treatment with PEMF in 8 weeks

SUMMARY:
PEMF (Pulsed Electro Magnetic Fields) therapy has been used to stimulate bone repair in non-union since the 1970s. This is an accepted use, which has been approved by the Food and Drug Administration in the US. The mode of action of PEMF is based on creating small electrical fields in tissue and thereby promoting healing. Besides it has been shown that PEMF enhance regeneration of nerve fibers exposed to a lesion For treatment of depression the PEMF equipment, which are provided by the company Re5 A/S, consists of a 220 V impulse generator that creates electrical impulses and an applicator which consists of an electrical cable connected to a helmet on which there are 7 electrical coils on the inside. In comparison with the rTMS (Transcranial Magnetic Stimulation) equipment, which uses stimuli approaching neuronal firing level, the PEMF fields in human is very much lower.

DETAILED DESCRIPTION:
Applied to cells PEMF have a stimulatory effect on intracellular tyrosine kinase activity, especially the Src family. The Src family upregulate NMDAR (N-methyl-D-aspartate) subtype of glutamate receptor thereby gating the production of NMDAR-dependent synaptic potentiation that are vital for processes that underlie physiological and pathological plasticity in the brain. Dysregulation of fibroblast growth factor receptors in frontal cortical regions of the brain seem to be associated with depression. The fibroblast growth factors are highly dependent on the activity of the Src family.

For treatment of depression the PEMF equipment, which are provided by the company Re5 A/S, consists of a 220 V impulse generator that creates electrical impulses and an applicator which consists of an electrical cable connected to a helmet on which there are 7 electrical coils on the inside. In comparison with the rTMS equipment, which uses stimuli approaching neuronal firing level, the PEMF fields in human are very much lower.

PEMF treatment involves placing the treatment helmet on the head and connecting it to a power source (220 V), which leads to induction of a pulsating magnetic field. The treatment was given for 30 min once or twice daily for 8 weeks. Participants are awake during these treatments and sit in a chair where they can read or eat. Pilot data demonstrates that the treatment can give mild transient nausea. No other side effects have been observed.

ELIGIBILITY:
Inclusion Criteria:

* Treatment resistant depression is defined as treatment with at least two antidepressants from different classes in an optimal dose and with sufficient duration (at least 8 weeks).
* A score on HamD17 above 17.
* Antidepressant medication must not have been changed 4 weeks before inclusion.

Exclusion Criteria:

A Ham-D17 item 3 at 2 or more (suicidal risk increased) A moderate manic condition (MAS-M above 14) The participant must not be under some sort of restrictions Pregnancy Severe personality disorders Psychotic mental disorders Brain diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Scale (HAM-D17) | 8 weeks
  HamD17 scale

SECONDARY OUTCOMES:
Life Quality | 8 weeks
  WHO-5 scale
Side effects | 8 weeks
  Prise scale
Response and remission | 8 weeks
  HamD17 scale

CONTACTS AND LOCATIONS:
Overall Officials: Erik R. Larsen, MD, Principal Investigator — Institute of Clinical Research, Research Unit of Psychiatry, University of Southern Denmark
Locations (1):
- Department of Psychiatry, Psychiatry in the Region of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Publication in Peer-Reviewed Journals Participation in Congresses
Supporting Information: Study Protocol
Time Frame: Planned to be published in 2018